CLINICAL TRIAL: NCT05979506
Title: Evaluate the Evolution of Cutaneous Discomfort of the Body and Scalp After 3 Wraps, in Patients With Moderate to Very Severe Hereditary Ichthyosis
Brief Title: Evaluate the Evolution of Body and Scalp Skin Discomfort in Patients With Hereditary Ichthyosis After Wraps (EnvelopIchtyose)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/21/0341
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Ichthyosis Inherited
Keywords: Ichthyosis; inherited; wraps; skin scales; cutaneous abnormalities
MeSH Terms: conditions — Ichthyosis

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, multicenter (Toulouse - Bordeaux - Paris Necker), comparative (baseline vs. short and medium term)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wraps (body and feet) as well as scalp care (Experimental): The skin care consisting of wraps (body and feet) and scalp care, will be carried out consecutively over 3 days, in the hospital (outpatient or in day/traditional hospitalization).
  Interventions: Procedure: Cutaneous wraps

INTERVENTIONS:
Procedure: Cutaneous wraps — The topical treatment that will be used in this study are:
  * For the body, an emollient cream with a high lipid content: Cold cream
  * For the scalp and feet, an emollient preparation with keratolytic action: 10% or 30% urea, depending on the scalp and feet damage
  Each of the 3 treatments (body, scalp and feet) will be carried out as follows:
  * Application of different topicals all over the body and face, after taking a lukewarm therapeutic bath of 20 minutes
  * Occlusion by "wrapping" the patient in a plastic film, then covering with a blanket
  * After 1 hour, the unabsorbed excess cream is removed with a towel

SUMMARY:
Ichthyosis is a group of rare and chronic genetic diseases beginning at birth, in which the patient's skin is covered with scales of variable appearance and severity. This disease is disabling. The treatment is symptomatic and is based on the daily application of moisturizing creams with a high lipid content. Nevertheless, the effectiveness of these treatments is limited and are considered very painful by the patients. Wraps are local treatments carried out by specialized nurses and which consist in, following a therapeutic bath, applying a large quantity of cream to the whole body, followed by an occlusion. This type of care is simple to perform, but requires nursing expertise, to date, it is not carried out in standard practice in France, which is why the investigateur wish to evaluate the effect of wraps on different parameters reflecting the skin condition in the short and medium term.

DETAILED DESCRIPTION:
Ichthyosis is a group of rare and chronic genetic diseases beginning at birth, in which the patient's skin is covered with scales of variable appearance and severity. There are 2 distinct typical profiles: patients with thick scales without erythroderma and patients with finer scales on an erythrodermic background. This disease is disabling, in particular due to sensations of pruritus, skin pain and the possible presence of associated extra-cutaneous abnormalities. The treatment is symptomatic and is based on the daily application of moisturizing creams with a high lipid content for better effectiveness, keratolytic creams, and for severe forms, oral retinoids may be necessary. The creams improve the condition of the skin and reduce the sensations of skin discomfort, pain and pruritus, nevertheless, the effectiveness of these treatments is limited and are considered very painful by the patients.

Wraps are local treatments carried out by specialized nurses and which consist in, following a therapeutic bath, applying a large quantity of cream to the whole body, followed by an occlusion. The type of cream is adapted to the area of application: thus, an emollient cream is used for the body; a cream enriched with keratolytic active ingredients is used for the feet in the event of hyperkeratosis, and an emollient cream possibly enriched with keratolytic active ingredients is used for the scalp, followed by an exposure time under a steam helmet to remove scales. This type of care is simple to perform, but requires nursing expertise, to date, it is not carried out in standard practice in France, except in the centers of Toulouse, Bordeaux and Necker and at the thermal cure of Avène-les-Bains. However, the interest of such a treatment has never been evaluated independently, which is why in this study the investigators want to evaluate the effect of carrying out a daily treatment over 3 consecutive days, on different parameters reflecting the skin condition in the short and medium term

ELIGIBILITY:
Inclusion Criteria:

* Patient with hereditary ichthyosis regardless of the clinical form
* Patient with a scaling or erythema score > 6/16
* Patient with a skin discomfort score > 3/10
* Patient having given written, free and informed consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient with a skin disease other than ichthyosis
* Patient having modified his treatments for ichthyosis in the month preceding inclusion
* Patient with known intolerance or allergy to one of the topicals used in the study
* Patient unable to complete the study questionnaires
* Patient under a protection regime

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Skin discomfort Analogue Visual Scale (AVS) | day 11
  Percentage of patients showing a reduction of at least 3 points of their skin discomfort in the entire body, measured with the AVS scale (0-10) of cutaneous discomfort between baseline and 11 days after treatment

SECONDARY OUTCOMES:
Reduction of skin discomfort - day 4 | day 4
  Percentage of patients showing a reduction of at least 3 points of their skin discomfort in the entire body, measured with the Analogue Visual Scale (AVS) (0-10) of cutaneous discomfort between baseline and day 4
Reduction of skin discomfort - day 30 | day 30
  Percentage of patients showing a reduction of at least 3 points of their skin discomfort in the entire body, measured with the Analogue Visual Scale (AVS) (0-10) of cutaneous discomfort between baseline and day 30
Variation of erythema and scales severity - VIIS | day 4
  Variation of erythema and scales severity judged by :
  - Their intensity, measured with the Visual Index for Ichthyosis Severity (VIIS)
Variation of erythema and scales severity | day 4
  Variation of erythema and scales severity judged by :
  -Their extent, measured with the scores A and B of the Specific Clinical Ichthyosis Score
Cutaneous pain - day 4 | day 4
  Variation of pain assessed by the Analogue Visual Scale (0-10) of skin pain
pruritus - day 4 | day 4
  Variation of pruritus assessed by the Analogue Visual Scale (0-10)
sweating - day 4 | day 4
  Variation of sweating assessed by the Analogue Visual Scale (0-10)
Cutaneous pain - day 11 | day 11
  Variation of pain assessed by the Analogue Visual scale (0-10) of skin pain
pruritus - day 11 | day 11
  Variation of pruritus assessed by the Analogue Visual scale (0-10)
sweating - day 11 | day 11
  Variation of sweating assessed by the Analogue Visual Scale scale (0-10)
Cutaneous pain - day 30 | day 30
  Variation of pain assessed by the Analogue Visual Scale (0-10) of skin pain
pruritus - day 30 | day 30
  Variation of pruritus assessed by the Analogue Visual Scale scale (0-10)
sweating - day 30 | day 30
  Variation of sweating assessed by the Analogue Visual Scale (0-10)
Feet and scalp discomfort - day 4 | day 4
  Percentage of patients showing a reduction of at least 3 points of their skin discomfort in the feet and scalp, measured with the Analogue Visual Scale (0-10) of cutaneous discomfort
Feet and scalp discomfort - day 11 | day 11
  Percentage of patients showing a reduction of at least 3 points of their skin discomfort in the feet and scalp, measured with the Analogue Visual Scale (0-10) of cutaneous discomfort
Feet and scalp discomfort - day 30 | day 30
  Percentage of patients showing a reduction of at least 3 points of their skin discomfort in the feet and scalp, measured with the Analogue Visual Scale (0-10) of cutaneous discomfort
32-item Ichthyosis Quality of Life questionnaire (IQoL-32) | 30 days after treatment
  Variation of patient's quality of life, measured by the ichthyosis specific quality of life questionnaire (IQoL-32)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie TRANIER, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No